CLINICAL TRIAL: NCT03984825
Title: The Effect of Coadministration of GSK3640254 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel in Healthy Female Subjects
Brief Title: Effect of GSK3640254 on the Pharmacokinetics of a Combination Oral Contraceptive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208135
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: HIV Infections
Keywords: GSK3640254; ethinyl estradiol; levonorgestrel; oral contraceptive; drug-drug interaction
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Portia followed by Portia co-administered with GSK3640254 (Experimental): Subjects will be administered Portia (0.03 mg EE/0.15 mg LNG) once daily on Days -3 to -1 during run-in period and on Days 1 to 10 in treatment period A. Subjects will then receive Portia (0.03 mg EE/0.15 mg LNG) co-administered with GSK3640254 200 mg once daily on Days 11 to 21 in treatment period B.
  Interventions: Drug: GSK3640254; Drug: Portia

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 will be available as a 100 mg capsule. Subjects will be administered 200 mg GSK3640254 once daily via the oral route on Days 11 to 21.
Drug: Portia — Portia will be available in the form of tablets containing 0.03 mg ethinyl estradiol and 0.15 mg levonorgestrel.

SUMMARY:
This is an open-label, single-sequence, 1-way drug-drug interaction study to investigate the effect of GSK3640254 on the pharmacokinetics of a combination oral contraceptive containing ethinyl estradiol (EE) and levonorgestrel (LNG). Effective contraception for women infected with human immunodeficiency virus (HIV) is important in the prevention of unplanned pregnancies. The study will consist of a screening period of 28 days, check-in (Day -4), a run-in period and a treatment period. During the run-in period, subjects will be administered Portia® (0.03 milligrams [mg] EE/0.15 mg LNG) once daily on Days -3 to -1. Subjects will then be administered Portia once daily on Days 1 to 10 of treatment period A followed by administration of Portia once daily along with GSK3640254 200 mg on Days 11 to 21 of treatment period B. The duration of the study is approximately 8 weeks, including Screening and Run-in. Portia is a registered trademark of Teva Pharmaceuticals USA.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Subjects who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Body weight >=45.0 kilograms (kg) (99 pounds [lbs]) and body mass index (BMI) within the range 18.5 to 31.0 kilograms per meter square (kg/m^2) (inclusive).
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female subjects will be included.
* Subject must not be pregnant or breastfeeding.
* Subject is a woman of childbearing potential (WOCBP) with intact ovarian function, as determined by medical history. Subjects must use Portia for the duration of the run-in and treatment periods.
* WOCBP must have been on an acceptable form of contraceptive for at least 28 days prior to start of study intervention. Acceptable forms of contraception prior to study intervention include the following: Intrauterine device or intrauterine system; Combined estrogen and progestogen oral contraceptive; Contraceptive vaginal ring; Percutaneous contraceptive patches (if used, the patch must be removed during study participation); Bilateral tubal occlusion; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. The documentation on male sterility can come from the site personnel's review of subject's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner.; Sexual abstinence.
* Subjects who have been on a stable regimen of an oral contraceptive for at least 3 consecutive months must be without evidence of breakthrough bleeding or spotting.
* Subjects who have been taking oral contraceptives should continue their current regimen until check-in to the clinic for the run-in period. Subjects not currently taking an oral contraceptive are eligible, provided all other eligibility criteria are met.
* Subjects may proceed to the treatment period provided the toxicity profile during the run-in period with Portia is acceptable in the opinion of the investigator.
* Subjects must agree to use an additional method of contraception from the following list of contraceptive methods for the run-in period, treatment period, and for 28 days after the last dose of study intervention: Non hormonal Intrauterine device; Bilateral tubal occlusion; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. The documentation on male sterility can come from the site personnel's review of subject's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner.; Sexual abstinence. For the 28 days after study exit, women may resume oral contraceptives but double barrier methods (a combination of male condom with either cervical cap, diaphragm, or sponge with spermicide) must be used in addition.
* Women of childbearing potential must have a negative highly sensitive serum pregnancy test on Day -4 and Day -1.
* Additional requirements for pregnancy testing during and after study intervention as outlined in protocol.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and protocol.

Exclusion Criteria:

* History of jaundice associated with taking oral contraceptives or with pregnancy.
* History of clinically significant irregular bleeding while taking oral contraceptives.
* History of past deep venous thrombosis, pulmonary embolism, stroke, transient ischemic attack, phlebitis, or migraine headaches with prolonged aura.
* History of cerebrovascular or coronary artery disease.
* History of retinal vascular lesions.
* History of carcinoma of the breast, endometrium, or other known estrogen-dependent neoplasia.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastrointestinal (GI) anatomy or motility (e.g., gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs or render the subject unable to take oral study intervention.
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Subjects with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Healthcare/GlaxoSmithKline (GSK) Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the subject's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the subject.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention AND positive on reflex to hepatitis C ribonucleic acid (RNA).
* Positive HIV-1 and -2 antigen/antibody immunoassay at Screening.
* ALT >1.5 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides, etc), and ALT (described above), will exclude a subject from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or nonprescription drugs including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study (acetaminophen/paracetamol at doses of <=2 grams/day and hydrocortisone cream 1% are permitted for use any time during the study).
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia Suicide Severity Rating Scale (C-SSRS).
* Any significant arrhythmia or ECG finding (e.g., symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, second-degree atrioventricular block Mobitz Type II, or third-degree atrioventricular block) which, in the opinion of the investigator or ViiV Healthcare/GSK Medical Monitor, will interfere with the safety for the individual subject.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): heart rate-<50 or >100 beats per minute and QTcF->450 milliseconds.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units. One unit is equivalent to 8 g of alcohol: a half-pint (equivalent to 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Unable to refrain from tobacco- or nicotine-containing within 3 months prior to Screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, open-label, fixed-sequence, 1-way drug-drug interaction (DDI) study to assess the Pharmacokinetic (PK), pharmacodynamic (PD), safety, and tolerability of GSK3640254 and an oral contraceptive containing Ethinyl estradiol/Levonorgestrel (EE/LNG, Portia) when administered alone and in combination in healthy female participants.
Pre-assignment Details: A total of 23 participants were enrolled in the study
Groups:
- Portia Followed by Portia + GSK3640254: Participants in Run-in period received Portia (0.03 milligram [mg] EE/0.15 mg LNG) once daily (QD) on Day -3 through Day -1. Participants in Treatment Period 1 received Portia (0.3 mg EE/ 0.15 mg LNG) QD on Day 1 through Day 10. In Treatment Period 2 participants received Portia QD co-administered with GSK3640254 200 mg QD on Day 11 through Day 21. There was no washout period between two periods.
Period: Run-in Period (Day -3 to -1)
Arm/Group | Portia Followed by Portia + GSK3640254
Started | 23
Completed | 23
Not Completed | 0
Period: Treatment Period 1 (Day 1 to 10)
Arm/Group | Portia Followed by Portia + GSK3640254
Started | 23
Completed | 21
Not Completed | 2
Not completed — Sponsor decision | 2
Period: Treatment Period 2 (Day 11 to 21)
Arm/Group | Portia Followed by Portia + GSK3640254
Started | 21
Completed | 17
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Portia Followed by Portia + GSK3640254
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.7 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian-Central/South Asian Heritage | 1
  Black or African American | 12
  White | 9

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Time 0 to the End of the Dosing Interval at Steady State (AUC [0-tau]) of EE
Description: Blood samples were collected at indicated time points for the analysis of AUC (0-tau) of EE. PK parameters were calculated by standard non-compartmental analysis. The PK population included all participants who underwent plasma PK sampling and had evaluable PK parameters estimated.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picograms per milliliter
Groups:
- Portia (0.3 mg EE/ 0.15 mg LNG): Participants in period 1 received Portia (0.3 mg of EE and 0.15 mg LNG) QD on Day 1 through Day 10.
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Hour*picograms per milliliter | 748.7 (25.2)

2. Primary Outcome: Period 2: AUC (0-tau) of EE
Description: Blood samples were collected at indicated time points for the analysis of AUC (0-tau) of EE. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 and 24 hours post dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picograms per milliliter
Groups:
- Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254: Participants in treatment period 2 were co-administered with GSK3640254 200 mg QD along with Portia from Day 11 through Day 21.
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hour*picograms per milliliter | 735.8 (23.6)

3. Primary Outcome: Period 1:AUC (0-tau) of LNG
Description: Blood samples were collected at indicated time points for the analysis of AUC (0-tau) of LNG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Hour*picograms per milliliter | 68682.4 (40.3)

4. Primary Outcome: Period 2: AUC (0-tau) of LNG
Description: as for outcome 3
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 and 24 hours post dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hour*picograms per milliliter | 75412.0 (40.7)

5. Primary Outcome: Period 1: Maximum Observed Concentration (Cmax) and Plasma Concentration at the End of the Dosing Interval (Ctau) of EE
Description: Blood samples were collected at indicated time points for the analysis of Cmax and Ctau of EE. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Picograms per milliliter
  Cmax | 70.01 (34.9)
  Ctau | 14.83 (32.1)

6. Primary Outcome: Period 2: Cmax and Ctau of EE
Description: as for outcome 5
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 and 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Picograms per milliliter
  Cmax | 68.47 (33.3)
  Ctau | 15.69 (27.8)

7. Primary Outcome: Period 1:Cmax and Ctau of LNG
Description: Blood samples were collected at indicated time points for the analysis of Cmax and Ctau of LNG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Picograms per milliliter
  Cmax | 5806 (39.3)
  Ctau | 1870 (49.0)

8. Primary Outcome: Period 2: Cmax and Ctau of LNG
Description: as for outcome 7
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 and 24 hours post dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Picograms per milliliter
  Cmax | 5948 (36.7)
  Ctau | 2163 (46.6)

9. Secondary Outcome: Period 1: Effect of GSK3640254 on PD of EE/LNG- Serum Progesterone Level
Description: Serum samples were collected for the analysis of progesterone concentration levels when GSK3640254 is co-administered with EE/LNG. PD concentration Population comprised of all participants who underwent plasma PD sampling and had evaluable PD assay results.
Time Frame: At Day 1 and Day 10
Population: PD concentration Population.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Nanomoles per liter
  Day 1 | 6.103 (5.0947)
  Day 10 | 4.410 (1.5370)

10. Secondary Outcome: Period 2: Effect of GSK3640254 on PD of EE/LNG- Serum Progesterone Level
Description: Serum samples were collected for the analysis progesterone concentration levels when GSK3640254 is co-administered with EE/LNG.
Time Frame: At Days 11, 21 and 22
Population: PD concentration Population. Only those participants with data available at specified time points has been presented (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Nanomoles per liter
  Day 11, n=21 | 3.906 (1.2178)
  Day 21, n=17: number analyzed (Participants) | 17
  Day 21, n=17 | 3.618 (0.9386)
  Day 22, n=17: number analyzed (Participants) | 17
  Day 22, n=17 | 3.988 (1.4316)

11. Secondary Outcome: Period 1: Absolute Values of Effect of GSK3640254 on Luteinizing Hormone (LH) and Follicle-stimulating Hormone (FSH)
Description: Serum samples were collected for the analysis of effect of GSK3640254 on LH and FSH.
Time Frame: At Day 1 and Day 10
Population: PD concentration Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
International units per liter
  LH, Day 1 | 9.500 (11.0104)
  LH, Day 10 | 2.747 (1.9554)
  FSH, Day 1 | 5.109 (3.7754)
  FSH, Day 10 | 2.215 (1.4567)

12. Secondary Outcome: Period 2: Absolute Values of Effect of GSK3640254 on LH and FSH
Description: Serum samples were collected for the analysis of effect of GSK3640254 on LH and FSH.
Time Frame: At Days 11, 21 and 22
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
International units per liter
  LH, Day 11, n=21 | 2.255 (1.6299)
  LH, Day 21, n=17: number analyzed (Participants) | 17
  LH, Day 21, n=17 | 1.202 (0.6667)
  LH, Day 22, n=17: number analyzed (Participants) | 17
  LH, Day 22, n=17 | 1.287 (0.8298)
  FSH, Day 11, n=21 | 2.162 (1.4388)
  FSH, Day 21, n=17: number analyzed (Participants) | 17
  FSH, Day 21, n=17 | 1.535 (0.8285)
  FSH, Day 22, n=17: number analyzed (Participants) | 17
  FSH, Day 22, n=17 | 1.638 (1.2380)

13. Secondary Outcome: Period 2: AUC (0-tau) of GSK3640254
Description: Blood samples were collected at indicated time points for the analysis of AUC (0-tau) of GSK3640254. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 21: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8 and 12 and 24 hours post dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hour*micrograms per milliliter | 30.22 (23.1)

14. Secondary Outcome: Period 2: Cmax and Ctau of GSK3640254
Description: Blood samples were collected at indicated time points for the analysis of Cmax and Ctau of GSK3640254. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 21: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8 and 12 and 24 hours post dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Micrograms per milliliter
  Cmax | 1.780 (30.4)
  Ctau | 0.9663 (27.1)

15. Secondary Outcome: Period 2: Apparent Terminal Phase Half-life (t1/2) of GSK3640254
Description: Blood samples were collected at indicated time points for the analysis of t1/2 of GSK3640254. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 21: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8 and 12 hours; Day 22: 24 hours; Day 23: 48 hours; Day 24: 72 hours and Day 25: 96 hours
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 14
Hours | 25.656 (19.1)

16. Secondary Outcome: Period 2: Time of Maximum Observed Concentration (Tmax) of GSK3640254
Description: Blood samples were collected at indicated time points for the analysis of Tmax of GSK3640254. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 21: Pre-dose, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8 and 12 and 24 hours post dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hours | 4.500 [3.50 to 24.00]

17. Secondary Outcome: Period 1: t1/2 of EE
Description: Blood samples were collected at indicated time points for the analysis of t1/2 of EE. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Hours | NA (NA) — Not applicable(NA) indicated t1/2 could not be calculated as we need atleast 3 timepoints after Cmax within same participant and this criteria was not fulfilled due to insufficient sampling(upto 24hours,which was less than 3times estimated half life)

18. Secondary Outcome: Period 2: t1/2 of EE
Description: as for outcome 17
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 22: 24 hours; Day 23: 48 hours and Day 24: 72 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hours | 20.215 (17.4)

19. Secondary Outcome: Period 1: Tmax of EE
Description: Blood samples were collected at indicated time points for the analysis of Tmax of EE. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Hours | 2.000 [1.00 to 4.00]

20. Secondary Outcome: Period 2: Tmax of EE
Description: as for outcome 19
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 22: 24 hours; Day 23: 48 hours and Day 24: 72 hours
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hours | 2.000 [1.00 to 4.00]

21. Secondary Outcome: Period 1: t1/2 of LNG
Description: Blood samples were collected at indicated time points for the analysis of t1/2 of LNG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Hours | NA (NA) — Not applicable(NA) indicated t1/2 could not be calculated as we need atleast 3 timepoints after Cmax within same participant and this criteria was not fulfilled due to insufficient sampling(upto 24hours,which was less than 3times estimated half life)

22. Secondary Outcome: Period 2: t1/2 of LNG
Description: as for outcome 21
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours; Day 22: 24 hours; Day 23: 48 hours and Day 24: 72 hours
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 4
Hours | 30.100 (4.2)

23. Secondary Outcome: Period 1: Tmax of LNG
Description: Blood samples were collected at indicated time points for the analysis of Tmax of LNG. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 10: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours and Day 11: 24 hours
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Hours | 2.000 [0.50 to 4.00]

24. Secondary Outcome: Period 2: Tmax of LNG
Description: as for outcome 23
Time Frame: Day 21: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 7, 12 hours; Day 22: 24 hours; Day 23: 48 hours and Day 24: 72 hours
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Hours | 2.000 [1.00 to 4.00]

25. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAE) (Treatment Period)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. Safety Population comprised of all participants who received at least one dose of study medication.
Time Frame: Up to Day 25
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG) | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 23 | 21
Participants
  Non-serious AE | 5 | 9
  SAE | 0 | 0

26. Secondary Outcome: Number of Participants With Non-SAEs and SAE (Run-in Period)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: From Day -3 to Day -1
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Portia - Run-in Period (Day -3 to Day -1): Participants in Run-in period received Portia (0.03 mg EE/0.15 mg LNG) QD on Day -3 through Day -1.
Arm/Group | Portia - Run-in Period (Day -3 to Day -1)
Number analyzed (Participants) | 23
Participants
  Non-serious AE | 0
  SAE | 0

27. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium and Blood Urea Nitrogen (BUN)
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including Glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and BUN. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Millimoles per liter
  Glucose | -0.217 (0.3567)
  Cholesterol | -0.153 (0.3219)
  Triglycerides | -0.049 (0.2231)
  Anion gap | 1.3 (1.66)
  Calcium | 0.039 (0.0626)
  Carbon dioxide | -1.8 (1.30)
  Chloride | 0.1 (1.82)
  Phosphate | -0.030 (0.1056)
  Potassium | -0.03 (0.343)
  Sodium | -0.3 (2.12)
  BUN | -0.180 (0.5956)

28. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium and BUN
Description: as for outcome 27
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Millimoles per liter
  Glucose, Day 21 | -0.141 (0.2553)
  Glucose, Day 24 | 0.084 (0.2043)
  Cholesterol, Day 21 | -0.161 (0.2891)
  Cholesterol, Day 24 | 0.075 (0.4580)
  Triglycerides, Day 21 | -0.008 (0.1524)
  Triglycerides, Day 24 | -0.066 (0.1786)
  Anion gap, Day 21 | -1.5 (1.12)
  Anion gap, Day 24 | -0.6 (1.80)
  Calcium, Day 21 | -0.034 (0.0546)
  Calcium, Day 24 | 0.000 (0.0643)
  Carbon dioxide, Day 21 | 0.7 (1.16)
  Carbon dioxide, Day 24 | 1.6 (0.87)
  Chloride, Day 21 | -0.6 (1.06)
  Chloride, Day 24 | 0.5 (1.33)
  Phosphate, Day 21 | -0.074 (0.1073)
  Phosphate, Day 24 | -0.064 (0.0878)
  Potassium, Day 21 | -0.06 (0.253)
  Potassium, Day 24 | -0.02 (0.235)
  Sodium, Day 21 | -1.2 (1.03)
  Sodium, Day 24 | 1.5 (1.66)
  BUN, Day 21 | -0.664 (0.5033)
  BUN, Day 24 | -0.568 (0.4591)

29. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameters: Plasma Albumin, Globulin and Protein
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including plasma albumin, globulin and protein. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Grams per liter
  Albumin | -0.1 (1.62)
  Globulin | 1.0 (1.60)
  Protein | 0.9 (2.94)

30. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameters: Plasma Albumin, Globulin and Protein
Description: as for outcome 29
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Grams per liter
  Albumin, Day 21 | -0.5 (1.46)
  Albumin, Day 24 | 0.1 (2.52)
  Globulin, Day 21 | -0.4 (1.54)
  Globulin, Day 24 | 0.8 (1.91)
  Protein, Day 21 | -0.9 (2.73)
  Protein, Day 24 | 0.9 (4.31)

31. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameters: Plasma Amylase and Lipase
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including plasma amylase and lipase. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Units per liter
  Amylase | -0.7 (7.83)
  Lipase | 2.1 (4.03)

32. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameters: Plasma Amylase and Lipase
Description: as for outcome 31
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Units per liter
  Amylase, Day 21 | 3.2 (6.03)
  Amylase, Day 24 | 5.2 (6.69)
  Lipase, Day 21 | 1.8 (3.77)
  Lipase, Day 24 | 1.6 (3.33)

33. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameters: Plasma Creatine Kinase, Lactate Dehydrogenase, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Gamma Glutamyl Transferase (GGT)
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including Plasma creatine kinase, lactate dehydrogenase, ALT, ALP, AST and GGT. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
International units per liter
  Creatine kinase | -3.6 (19.7)
  lactate dehydrogenase | 0.0 (11.76)
  ALT | 11.5 (24.80)
  ALP | -3.9 (5.89)
  AST | 3.6 (9.74)
  GGT | 1.7 (8.36)

34. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameters: Plasma Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST and GGT
Description: as for outcome 33
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Units per liter
  Creatine kinase, Day 21 | -1.6 (9.51)
  Creatine kinase, Day 24 | -1.7 (12.18)
  Lactate dehydrogenase, Day 21 | 4.2 (10.61)
  Lactate dehydrogenase, Day 24 | 8.4 (16.00)
  ALT, Day 21 | 25.7 (24.80)
  ALT, Day 24 | 34.5 (37.36)
  ALP, Day 21 | -1.1 (2.38)
  ALP, Day 24 | -1.9 (3.60)
  AST, Day 21 | 10.1 (9.97)
  AST, Day 24 | 12.6 (15.62)
  GGT, Day 21 | 0.0 (1.73)
  GGT, Day 24 | 0.1 (1.60)

35. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameters: Plasma Urate, Creatinine, Total Bilirubin and Direct Bilirubin
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including Plasma urate, creatinine, total bilirubin and direct bilirubin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Micromoles per liter
  Urate | -18.0 (19.09)
  Creatinine | 0.93 (3.079)
  Total bilirubin | -0.57 (1.638)
  Direct bilirubin | -0.21 (0.467)

36. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameters: Plasma Urate, Creatinine, Total Bilirubin and Direct Bilirubin
Description: as for outcome 35
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Micromoles per liter
  Urate, Day 21 | -45.2 (19.22)
  Urate, Day 24 | -34.7 (19.63)
  Creatinine, Day 21 | 0.52 (2.852)
  Creatinine, Day 24 | 1.29 (3.013)
  Total bilirubin, Day 21 | 0.08 (1.000)
  Total bilirubin, Day 24 | 0.12 (1.177)
  Direct bilirubin, Day 21 | 0.07 (0.214)
  Direct bilirubin, Day 24 | 0.15 (0.318)

37. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples were collected at indicated time points for the analysis of hematology parameters including Basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
10^9 cells per liter
  Basophils | 0.000 (0.0133)
  Eosinophils | 0.008 (0.0263)
  Leukocytes | -0.02 (0.867)
  Lymphocytes | 0.086 (0.2168)
  Monocytes | -0.012 (0.0760)
  Neutrophils | -0.103 (0.7505)
  Platelets | -1.6 (32.32)

38. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: as for outcome 37
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
10^9 cells per liter
  Basophils, Day 21 | 0.001 (0.0130)
  Basophils, Day 24 | 0.000 (0.0150)
  Eosinophils, Day 21 | 0.001 (0.0209)
  Eosinophils, Day 24 | -0.005 (0.0414)
  Leukocytes, Day 21 | -0.43 (0.905)
  Leukocytes, Day 24 | -0.88 (0.901)
  Lymphocytes, Day 21 | -0.095 (0.2468)
  Lymphocytes, Day 24 | -0.101 (0.1617)
  Monocytes, Day 21 | -0.045 (0.0609)
  Monocytes, Day 24 | -0.064 (0.0676)
  Neutrophils, Day 21 | -0.285 (0.7448)
  Neutrophils, Day 24 | -0.708 (0.7253)
  Platelets, Day 21 | 12.2 (31.07)
  Platelets, Day 24 | 6.8 (27.18)

39. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter erythrocytes mean corpuscular hemoglobin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Picograms | -0.09 (0.366)

40. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: as for outcome 39
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Picograms
  Day 21 | -0.51 (0.394)
  Day 24 | -0.10 (0.377)

41. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter erythrocytes mean corpuscular volume. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Femtoliters | -0.18 (0.657)

42. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: as for outcome 41
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Femtoliters
  Day 21 | -0.50 (0.516)
  Day 24 | 0.04 (0.818)

43. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter erythrocytes. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
10^12 cells per liter | -0.010 (0.1287)

44. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Erythrocytes
Description: as for outcome 43
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
10^12 cells per liter
  Day 21 | 0.106 (0.1093)
  Day 24 | 0.134 (0.1675)

45. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter hematocrit. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Proportion of red blood cells in blood | -0.0014 (0.01165)

46. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: as for outcome 45
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Proportion of red blood cells in blood
  Day 21 | 0.0071 (0.01046)
  Day 24 | 0.0118 (0.01711)

47. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter hemoglobin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Grams per liter | -0.7 (3.74)

48. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: as for outcome 47
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 17
Grams per liter
  Day 21 | 1.2 (3.63)
  Day 24 | 3.8 (5.45)

49. Secondary Outcome: Period 1: Change From Baseline in Urine Concentration: Urine Specific Gravity
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Ratio | 0.0023 (0.00922)

50. Secondary Outcome: Period 2: Change From Baseline in Urine Concentration: Urine Specific Gravity
Description: as for outcome 49
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population. Only those participants with data available at specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Ratio
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | -0.0028 (0.01150)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | -0.0021 (0.00888)

51. Secondary Outcome: Period 1: Change From Baseline in Urine Concentration: Urine Urobilinogen
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Micromoles per liter | 1.7666 (4.66388)

52. Secondary Outcome: Period 2: Change From Baseline in Urine Concentration: Urine Urobilinogen
Description: as for outcome 51
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Micromoles per liter
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 3.0098 (5.79402)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.0000 (4.78853)

53. Secondary Outcome: Period 1: Change From Baseline in Urine Concentration: Urine Potential of Hydrogen (pH)
Description: Urine samples were collected at indicated time points for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
pH | -0.22 (0.473)

54. Secondary Outcome: Period 2: Change From Baseline in Urine Concentration: Urine pH
Description: as for outcome 53
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
pH
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 0.39 (0.583)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.24 (0.400)

55. Secondary Outcome: Period 1: Change From Baseline in Electrocardiogram (ECG) Mean Heart Rate
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure heart rate. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Beats per minute | -0.8 (5.95)

56. Secondary Outcome: Period 2: Change From Baseline in ECG Mean Heart Rate
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure heart rate. Baseline is defined as the average of the triplicate predose assessments on Day 11. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 11, Pre-dose) and at Day 11: 2, 4, 6 hours, Day 15: 2, 4, 6 hours, Day 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Beats per minute
  Day 11: 2 hours, n=21 | 2.8 (5.17)
  Day 11: 4 hours, n=21 | -0.6 (4.79)
  Day 11: 6 hours, n=21 | 6.7 (5.44)
  Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  Day 15: 2 hours, n=18 | 3.8 (6.23)
  Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  Day 15: 4 hours, n=18 | 1.7 (8.01)
  Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  Day 15: 6 hours, n=18 | 3.1 (7.10)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 3.7 (6.24)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.6 (4.42)

57. Secondary Outcome: Period 1: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, Fridericia QT Correction Formula (QTcF) Interval, and Bazett QT Correction Formula (QTcB) Interval
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure PR interval, QRS duration, QT Interval, QTcF Interval and QTcB interval. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Milliseconds
  PR interval | 2.5 (8.65)
  QRS duration | 0.2 (5.01)
  QT interval | -3.0 (11.32)
  QTcF interval | -4.1 (8.18)
  QTcB interval | -4.6 (11.80)

58. Secondary Outcome: Period 2: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF and QTcB Interval
Description: as for outcome 56
Time Frame: Baseline (Day 11, Pre-dose) and at Day 11: 2, 4, 6 hours, Day 15: 2, 4, 6 hours, Day 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Milliseconds
  PR interval, Day 11: 2 hours, n=21 | 0.3 (7.99)
  PR interval, Day 11: 4 hours, n=21 | 1.9 (8.68)
  PR interval, Day 11: 6 hours, n=21 | -1.9 (9.45)
  PR interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  PR interval, Day 15: 2 hours, n=18 | -1.7 (11.37)
  PR interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  PR interval, Day 15: 4 hours, n=18 | -0.6 (10.03)
  PR interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  PR interval, Day 15: 6 hours, n=18 | -2.3 (7.99)
  PR interval, Day 21, n=18: number analyzed (Participants) | 18
  PR interval, Day 21, n=18 | 1.7 (7.37)
  PR interval, Day 24, n=17: number analyzed (Participants) | 17
  PR interval, Day 24, n=17 | 2.1 (7.89)
  QRS duration, Day 11: 2 hours, n=21 | -2.2 (3.78)
  QRS duration, Day 11: 4 hours, n=21 | -0.7 (4.51)
  QRS duration, Day 11: 6 hours, n=21 | -0.3 (4.33)
  QRS duration, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QRS duration, Day 15: 2 hours, n=18 | 0.2 (3.78)
  QRS duration, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QRS duration, Day 15: 4 hours, n=18 | 0.1 (3.39)
  QRS duration, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QRS duration, Day 15: 6 hours, n=18 | -0.9 (3.02)
  QRS duration, Day 21, n=18: number analyzed (Participants) | 18
  QRS duration, Day 21, n=18 | -0.4 (4.37)
  QRS duration, Day 24, n=17: number analyzed (Participants) | 17
  QRS duration, Day 24, n=17 | -0.4 (3.36)
  QT interval, Day 11: 2 hours, n=21 | -16.4 (8.23)
  QT interval, Day 11: 4 hours, n=21 | 2.3 (10.78)
  QT interval, Day 11: 6 hours, n=21 | -11.7 (10.22)
  QT interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QT interval, Day 15: 2 hours, n=18 | -10.3 (10.09)
  QT interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QT interval, Day 15: 4 hours, n=18 | -0.4 (15.78)
  QT interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QT interval, Day 15: 6 hours, n=18 | 2.2 (14.21)
  QT interval, Day 21, n=18: number analyzed (Participants) | 18
  QT interval, Day 21, n=18 | -7.4 (13.77)
  QT interval, Day 24, n=17: number analyzed (Participants) | 17
  QT interval, Day 24, n=17 | 0.1 (10.06)
  QTcF interval, Day 11: 2 hours, n=21 | -11.5 (8.78)
  QTcF interval, Day 11: 4 hours, n=21 | 1.4 (8.61)
  QTcF interval, Day 11: 6 hours, n=21 | 1.3 (7.68)
  QTcF interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 15: 2 hours, n=18 | -3.0 (6.15)
  QTcF interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 15: 4 hours, n=18 | 2.4 (9.71)
  QTcF interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 15: 6 hours, n=18 | 8.1 (9.07)
  QTcF interval, Day 21, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 21, n=18 | -0.3 (6.85)
  QTcF interval, Day 24, n=17: number analyzed (Participants) | 17
  QTcF interval, Day 24, n=17 | 1.4 (5.63)
  QTcB interval, Day 11: 2 hours, n=21 | -8.5 (13.11)
  QTcB interval, Day 11: 4 hours, n=21 | 1.0 (11.57)
  QTcB interval, Day 11: 6 hours, n=21 | 8.2 (11.84)
  QTcB interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 15: 2 hours, n=18 | 1.1 (11.25)
  QTcB interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 15: 4 hours, n=18 | 4.4 (15.09)
  QTcB interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 15: 6 hours, n=18 | 11.6 (12.41)
  QTcB interval, Day 21, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 21, n=18 | 3.6 (9.20)
  QTcB interval, Day 24, n=17: number analyzed (Participants) | 17
  QTcB interval, Day 24, n=17 | 2.5 (7.67)

59. Secondary Outcome: Period 1: Change From Baseline in Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline is defined as the average of the triplicate pre-dose assessments. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Millimeters of mercury
  SBP | -4.3 (9.45)
  DBP | -2.8 (7.84)

60. Secondary Outcome: Period 2: Change From Baseline in Vital Signs: SBP and DBP
Description: SBP and DBP were assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline is defined as as the average of the triplicate pre-dose assessments. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Millimeters of mercury
  SBP, Day 15, n=19: number analyzed (Participants) | 19
  SBP, Day 15, n=19 | 4.4 (6.51)
  SBP, Day 21, n=18: number analyzed (Participants) | 18
  SBP, Day 21, n=18 | 1.6 (4.89)
  SBP, Day 24, n=17: number analyzed (Participants) | 17
  SBP, Day 24, n=17 | 5.9 (6.95)
  DBP, Day 15, n=19: number analyzed (Participants) | 19
  DBP, Day 15, n=19 | 3.0 (5.08)
  DBP, Day 21, n=18: number analyzed (Participants) | 18
  DBP, Day 21, n=18 | 3.5 (3.38)
  DBP, Day 24, n=17: number analyzed (Participants) | 17
  DBP, Day 24, n=17 | 6.1 (5.27)

61. Secondary Outcome: Period 1: Change From Baseline in Pulse Rate
Description: Pulse rate was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline is defined as the average of the triplicate predose assessments. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Beats per minute | -0.2 (5.16)

62. Secondary Outcome: Period 2: Change From Baseline in Pulse Rate
Description: as for outcome 61
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Beats per minute
  Day 15, n=19: number analyzed (Participants) | 19
  Day 15, n=19 | 5.8 (5.06)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 1.8 (5.71)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.9 (5.48)

63. Secondary Outcome: Period 1: Change From Baseline in Respiratory Rate
Description: Respiratory rate was assessed at indicated time-points. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Breaths per minute | 2.3 (2.58)

64. Secondary Outcome: Period 2: Change From Baseline in Respiratory Rate
Description: as for outcome 63
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Breaths per minute
  Day 15, n=19: number analyzed (Participants) | 19
  Day 15, n=19 | 1.7 (3.07)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 0.6 (2.15)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.9 (3.61)

65. Secondary Outcome: Period 1: Change From Baseline in Temperature
Description: Temperature was assessed at indicated time-points. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Degree Celsius | 0.11 (0.452)

66. Secondary Outcome: Period 2: Change From Baseline in Temperature
Description: as for outcome 65
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Degree Celsius
  Day 15, n=19: number analyzed (Participants) | 19
  Day 15, n=19 | 0.15 (0.434)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 0.02 (0.537)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.25 (0.505)

67. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium and BUN
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including Glucose, cholesterol, triglycerides, anion gap, calcium, carbon dioxide, chloride, phosphate, potassium, sodium and BUN. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Millimoles per liter
  Glucose, Baseline | 5.104 (0.5019)
  Glucose, Day 10 | 4.887 (0.4616)
  Cholesterol, Baseline | 4.291 (0.9991)
  Cholesterol, Day 10 | 4.138 (0.8322)
  Triglycerides, Baseline | 1.084 (0.5437)
  Triglycerides, Day 10 | 1.035 (0.3940)
  Anion gap, Baseline | 9.9 (1.10)
  Anion gap, Day 10 | 11.2 (1.44)
  Calcium, Baseline | 2.310 (0.0652)
  Calcium, Day 10 | 2.349 (0.0593)
  Carbon dioxide, Baseline | 28.0 (1.17)
  Carbon dioxide, Day 10 | 26.2 (1.44)
  Chloride, Baseline | 103.4 (1.41)
  Chloride, Day 10 | 103.6 (1.83)
  Phosphate, Baseline | 1.165 (0.1000)
  Phosphate, Day 10 | 1.135 (0.0881)
  Potassium, Baseline | 4.23 (0.288)
  Potassium, Day 10 | 4.20 (0.265)
  Sodium, Baseline | 137.1 (1.24)
  Sodium, Day 10 | 136.7 (1.57)
  BUN, Baseline | 3.659 (0.7512)
  BUN, Day 10 | 3.478 (0.6738)

68. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Anion Gap, Calcium, Carbon Dioxide, Chloride, Phosphate, Potassium, Sodium and BUN
Description: as for outcome 67
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Millimoles per liter
  Glucose, Baseline, n=21 | 4.921 (0.4503)
  Glucose, Day 21, n=17: number analyzed (Participants) | 17
  Glucose, Day 21, n=17 | 4.769 (0.3922)
  Glucose, Day 24, n=17: number analyzed (Participants) | 17
  Glucose, Day 24, n=17 | 4.994 (0.3746)
  Cholesterol, Baseline, n=21 | 4.104 (0.8622)
  Cholesterol, Day 21, n=17: number analyzed (Participants) | 17
  Cholesterol, Day 21, n=17 | 3.857 (0.8765)
  Cholesterol, Day 24, n=17: number analyzed (Participants) | 17
  Cholesterol, Day 24, n=17 | 4.093 (1.0474)
  Triglycerides, Baseline, n=21 | 1.032 (0.4092)
  Triglycerides, Day 21, n=17: number analyzed (Participants) | 17
  Triglycerides, Day 21, n=17 | 1.080 (0.4505)
  Triglycerides, Day 24, n=17: number analyzed (Participants) | 17
  Triglycerides, Day 24, n=17 | 1.022 (0.5161)
  Anion gap, Baseline, n=21 | 11.2 (1.48)
  Anion gap, Day 21, n=17: number analyzed (Participants) | 17
  Anion gap, Day 21, n=17 | 9.6 (1.46)
  Anion gap, Day 24, n=17: number analyzed (Participants) | 17
  Anion gap, Day 24, n=17 | 10.5 (1.42)
  Calcium, Baseline, n=21 | 2.349 (0.0602)
  Calcium, Day 21, n=17: number analyzed (Participants) | 17
  Calcium, Day 21, n=17 | 2.314 (0.0706)
  Calcium, Day 24, n=17: number analyzed (Participants) | 17
  Calcium, Day 24, n=17 | 2.348 (0.0592)
  Carbon dioxide, Baseline, n=21 | 26.0 (1.43)
  Carbon dioxide, Day 21, n=17: number analyzed (Participants) | 17
  Carbon dioxide, Day 21, n=17 | 26.7 (1.57)
  Carbon dioxide, Day 24, n=17: number analyzed (Participants) | 17
  Carbon dioxide, Day 24, n=17 | 27.6 (1.33)
  Chloride, Baseline, n=21 | 103.7 (1.74)
  Chloride, Day 21, n=17: number analyzed (Participants) | 17
  Chloride, Day 21, n=17 | 103.0 (2.18)
  Chloride, Day 24, n=17: number analyzed (Participants) | 17
  Chloride, Day 24, n=17 | 104.1 (2.01)
  Phosphate, Baseline, n=21 | 1.139 (0.0819)
  Phosphate, Day 21, n=17: number analyzed (Participants) | 17
  Phosphate, Day 21, n=17 | 1.055 (0.0908)
  Phosphate, Day 24, n=17: number analyzed (Participants) | 17
  Phosphate, Day 24, n=17 | 1.065 (0.0818)
  Potassium, Baseline, n=21 | 4.18 (0.211)
  Potassium, Day 21, n=17: number analyzed (Participants) | 17
  Potassium, Day 21, n=17 | 4.12 (0.198)
  Potassium, Day 24, n=17: number analyzed (Participants) | 17
  Potassium, Day 24, n=17 | 4.16 (0.197)
  Sodium, Baseline, n=21 | 136.9 (1.39)
  Sodium, Day 21, n=17: number analyzed (Participants) | 17
  Sodium, Day 21, n=17 | 135.4 (1.46)
  Sodium, Day 24, n=17: number analyzed (Participants) | 17
  Sodium, Day 24, n=17 | 138.1 (1.56)
  BUN, Baseline, n=21 | 3.458 (0.6189)
  BUN, Day 21, n=17: number analyzed (Participants) | 17
  BUN, Day 21, n=17 | 2.756 (0.4593)
  BUN, Day 24, n=17: number analyzed (Participants) | 17
  BUN, Day 24, n=17 | 2.853 (0.5406)

69. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameters: Plasma Albumin, Globulin and Protein
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including plasma albumin, globulin and protein. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Grams per liter
  Albumin, Baseline | 42.0 (2.29)
  Albumin, Day 10 | 42.0 (2.16)
  Globulin, Baseline | 28.8 (2.57)
  Globulin, Day 10 | 29.8 (2.93)
  Protein, Baseline | 70.9 (4.06)
  Protein, Day 10 | 71.8 (4.25)

70. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameters: Plasma Albumin, Globulin and Protein
Description: as for outcome 69
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Grams per liter
  Albumin, Baseline, n=21 | 41.9 (2.21)
  Albumin, Day 21, n=17: number analyzed (Participants) | 17
  Albumin, Day 21, n=17 | 41.4 (1.62)
  Albumin, Day 24, n=17: number analyzed (Participants) | 17
  Albumin, Day 24, n=17 | 42.0 (2.12)
  Globulin, Baseline, n=21 | 29.7 (2.99)
  Globulin, Day 21, n=17: number analyzed (Participants) | 17
  Globulin, Day 21, n=17 | 29.2 (2.70)
  Globulin, Day 24, n=17: number analyzed (Participants) | 17
  Globulin, Day 24, n=17 | 30.4 (2.50)
  Protein, Baseline, n=21 | 71.6 (4.40)
  Protein, Day 21, n=17: number analyzed (Participants) | 17
  Protein, Day 21, n=17 | 70.5 (3.68)
  Protein, Day 24, n=17: number analyzed (Participants) | 17
  Protein, Day 24, n=17 | 72.4 (3.97)

71. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameters: Plasma Amylase and Lipase
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including plasma amylase and lipase. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Units per liter
  Amylase, Baseline | 49.4 (18.77)
  Amylase, Day 10 | 48.7 (16.34)
  Lipase, Baseline | 18.8 (9.25)
  Lipase, Day 10 | 20.9 (8.47)

72. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameters: Plasma Amylase and Lipase
Description: as for outcome 71
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Units per liter
  Amylase, Baseline, n=21 | 47.8 (16.79)
  Amylase, Day 21, n=17: number analyzed (Participants) | 17
  Amylase, Day 21, n=17 | 47.1 (17.93)
  Amylase, Day 24, n=17: number analyzed (Participants) | 17
  Amylase, Day 24, n=17 | 49.2 (18.38)
  Lipase, Baseline, n=21 | 20.7 (8.83)
  Lipase, Day 21, n=17: number analyzed (Participants) | 17
  Lipase, Day 21, n=17 | 20.5 (7.40)
  Lipase, Day 24, n=17: number analyzed (Participants) | 17
  Lipase, Day 24, n=17 | 20.4 (8.16)

73. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameters: Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST and GGT
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including creatine kinase, lactate dehydrogenase, ALT, ALP, AST and GGT. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
International units per liter
  Creatine kinase, Baseline | 74.1 (25.37)
  Creatine kinase, Day 10 | 70.5 (22.43)
  Lactate dehydrogenase, Baseline | 122.7 (21.78)
  Lactate dehydrogenase, Day 10 | 122.7 (21.19)
  ALT, Baseline | 12.4 (6.45)
  ALT, Day 10 | 23.9 (24.34)
  ALP, Baseline | 49.6 (12.00)
  ALP, Day 10 | 45.7 (11.64)
  AST, Baseline | 14.2 (2.79)
  AST, Day 10 | 17.7 (9.26)
  GGT, Baseline | 14.9 (5.62)
  GGT, Day 10 | 16.7 (11.48)

74. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameters: Plasma Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST and GGT
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including Plasma creatine kinase, lactate dehydrogenase, ALT, ALP, AST and GGT. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
International units per liter
  Creatine kinase, Baseline, n=21 | 70.3 (23.37)
  Creatine kinase, Day 21, n=17: number analyzed (Participants) | 17
  Creatine kinase, Day 21, n=17 | 69.4 (23.62)
  Creatine kinase, Day 24, n=17: number analyzed (Participants) | 17
  Creatine kinase, Day 24, n=17 | 69.3 (22.46)
  Lactate dehydrogenase, Baseline, n=21 | 123.3 (21.96)
  Lactate dehydrogenase, Day 21, n=17: number analyzed (Participants) | 17
  Lactate dehydrogenase, Day 21, n=17 | 125.9 (24.85)
  Lactate dehydrogenase, Day 24, n=17: number analyzed (Participants) | 17
  Lactate dehydrogenase, Day 24, n=17 | 130.1 (27.63)
  ALT, Baseline, n=21 | 25.7 (27.34)
  ALT, Day 21, n=17: number analyzed (Participants) | 17
  ALT, Day 21, n=17 | 42.2 (32.02)
  ALT, Day 24, n=17: number analyzed (Participants) | 17
  ALT, Day 24, n=17 | 51.1 (45.07)
  ALP, Baseline, n=21 | 44.9 (10.91)
  ALP, Day 21, n=17: number analyzed (Participants) | 17
  ALP, Day 21, n=17 | 43.5 (10.46)
  ALP, Day 24, n=17: number analyzed (Participants) | 17
  ALP, Day 24, n=17 | 42.6 (10.10)
  AST, Baseline, n=21 | 17.7 (9.05)
  AST, Day 21, n=17: number analyzed (Participants) | 17
  AST, Day 21, n=17 | 25.4 (14.55)
  AST, Day 24, n=17: number analyzed (Participants) | 17
  AST, Day 24, n=17 | 27.9 (20.07)
  GGT, Baseline, n=21 | 16.4 (11.60)
  GGT, Day 21, n=17: number analyzed (Participants) | 17
  GGT, Day 21, n=17 | 13.0 (4.53)
  GGT, Day 24, n=17: number analyzed (Participants) | 17
  GGT, Day 24, n=17 | 13.1 (4.45)

75. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameters: Urate, Creatinine, Total Bilirubin and Direct Bilirubin
Description: Blood samples were collected at indicated time points for the analysis of clinical chemistry parameters including Plasma urate, creatinine, total bilirubin and direct bilirubin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Micromoles per liter
  Urate, Baseline | 260.4 (46.10)
  Urate, Day 10 | 242.4 (46.30)
  Creatinine, Baseline | 67.75 (8.763)
  Creatinine, Day 10 | 68.68 (9.846)
  Total bilirubin, Baseline | 8.35 (3.847)
  Total bilirubin, Day 10 | 7.79 (3.480)
  Direct bilirubin, Baseline | 1.88 (0.871)
  Direct bilirubin, Day 10 | 1.67 (0.701)

76. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameters: Plasma Urate, Creatinine, Total Bilirubin and Direct Bilirubin
Description: as for outcome 75
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Micromoles per liter
  Urate, Baseline, n=21 | 240.3 (43.74)
  Urate, Day 21, n=17: number analyzed (Participants) | 17
  Urate, Day 21, n=17 | 194.5 (35.17)
  Urate, Day 24, n=17: number analyzed (Participants) | 17
  Urate, Day 24, n=17 | 205.1 (39.09)
  Creatinine, Baseline, n=21 | 68.62 (10.637)
  Creatinine, Day 21, n=17: number analyzed (Participants) | 17
  Creatinine, Day 21, n=17 | 66.92 (6.770)
  Creatinine, Day 24, n=17: number analyzed (Participants) | 17
  Creatinine, Day 24, n=17 | 67.70 (7.456)
  Total bilirubin, Baseline, n=21 | 7.98 (3.563)
  Total bilirubin, Day 21, n=17: number analyzed (Participants) | 17
  Total bilirubin, Day 21, n=17 | 6.94 (1.600)
  Total bilirubin, Day 24, n=17: number analyzed (Participants) | 17
  Total bilirubin, Day 24, n=17 | 6.99 (2.323)
  Direct bilirubin, Baseline, n=21 | 1.72 (0.699)
  Direct bilirubin, Day 21, n=17: number analyzed (Participants) | 17
  Direct bilirubin, Day 21, n=17 | 1.56 (0.498)
  Direct bilirubin, Day 24, n=17: number analyzed (Participants) | 17
  Direct bilirubin, Day 24, n=17 | 1.64 (0.592)

77. Secondary Outcome: Period 1: Absolute Values of Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples were collected at indicated time points for the analysis of hematology parameters including Basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
10^9 cells per liter
  Basophils, Baseline | 0.038 (0.0239)
  Basophils, Day 10 | 0.038 (0.0177)
  Eosinophils, Baseline | 0.103 (0.0555)
  Eosinophils, Day 10 | 0.111 (0.0606)
  Leukocytes, Baseline | 6.23 (1.626)
  Leukocytes, Day 10 | 6.21 (1.329)
  Lymphocytes, Baseline | 1.730 (0.3832)
  Lymphocytes, Day 10 | 1.816 (0.3399)
  Monocytes, Baseline | 0.460 (0.1238)
  Monocytes, Day 10 | 0.448 (0.1144)
  Neutrophils, Baseline | 3.905 (1.2865)
  Neutrophils, Day 10 | 3.802 (1.1472)
  Platelets, Baseline | 284.4 (36.78)
  Platelets, Day 10 | 282.8 (45.94)

78. Secondary Outcome: Period 2: Absolute Values of Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: as for outcome 77
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
10^9 cells per liter
  Basophils, Baseline, n=21 | 0.039 (0.0184)
  Basophils, Day 21, n=17: number analyzed (Participants) | 17
  Basophils, Day 21, n=17 | 0.039 (0.0183)
  Basophils, Day 24, n=17: number analyzed (Participants) | 17
  Basophils, Day 24, n=17 | 0.038 (0.0142)
  Eosinophils, Baseline, n=21 | 0.115 (0.0622)
  Eosinophils, Day 21, n=17: number analyzed (Participants) | 17
  Eosinophils, Day 21, n=17 | 0.118 (0.0631)
  Eosinophils, Day 24, n=17: number analyzed (Participants) | 17
  Eosinophils, Day 24, n=17 | 0.112 (0.0645)
  Leukocytes, Baseline, n=21 | 6.20 (1.391)
  Leukocytes, Day 21, n=17: number analyzed (Participants) | 17
  Leukocytes, Day 21, n=17 | 5.86 (1.183)
  Leukocytes, Day 24, n=17: number analyzed (Participants) | 17
  Leukocytes, Day 24, n=17 | 5.41 (1.080)
  Lymphocytes, Baseline, n=21 | 1.790 (0.3089)
  Lymphocytes, Day 21, n=17: number analyzed (Participants) | 17
  Lymphocytes, Day 21, n=17 | 1.715 (0.3349)
  Lymphocytes, Day 24, n=17: number analyzed (Participants) | 17
  Lymphocytes, Day 24, n=17 | 1.710 (0.2207)
  Monocytes, Baseline, n=21 | 0.446 (0.1186)
  Monocytes, Day 21, n=17: number analyzed (Participants) | 17
  Monocytes, Day 21, n=17 | 0.409 (0.0942)
  Monocytes, Day 24, n=17: number analyzed (Participants) | 17
  Monocytes, Day 24, n=17 | 0.391 (0.0924)
  Neutrophils, Baseline, n=21 | 3.811 (1.2013)
  Neutrophils, Day 21, n=17: number analyzed (Participants) | 17
  Neutrophils, Day 21, n=17 | 3.587 (1.0893)
  Neutrophils, Day 24, n=17: number analyzed (Participants) | 17
  Neutrophils, Day 24, n=17 | 3.165 (0.9633)
  Platelets, Baseline, n=21 | 282.2 (46.73)
  Platelets, Day 21, n=17: number analyzed (Participants) | 17
  Platelets, Day 21, n=17 | 296.8 (50.45)
  Platelets, Day 24, n=17: number analyzed (Participants) | 17
  Platelets, Day 24, n=17 | 291.4 (42.75)

79. Secondary Outcome: Period 1: Absolute Values of Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter erythrocytes mean corpuscular hemoglobin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Picograms
  Baseline | 29.70 (2.010)
  Day 10 | 29.62 (2.228)

80. Secondary Outcome: Period 2: Absolute Values of Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: as for outcome 79
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Picograms
  Baseline, n=21 | 29.92 (2.068)
  Day 21, n=17: number analyzed (Participants) | 17
  Day 21, n=17 | 29.72 (1.779)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 30.12 (1.867)

81. Secondary Outcome: Period 1: Absolute Values of Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter erythrocytes mean corpuscular volume. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Femtoliters
  Baseline | 87.83 (5.060)
  Day 10 | 87.65 (4.991)

82. Secondary Outcome: Period 2: Absolute Values of Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: as for outcome 81
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Femtoliters
  Baseline, n=21 | 88.16 (4.889)
  Day 21, n=17: number analyzed (Participants) | 17
  Day 21, n=17 | 88.39 (4.293)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 88.92 (4.278)

83. Secondary Outcome: Period 1: Absolute Values of Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter erythrocytes. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
10^12 cells per liter
  Baseline | 4.316 (0.3113)
  Day 10 | 4.306 (0.3008)

84. Secondary Outcome: Period 2: Absolute Values of Hematology Parameter: Erythrocytes
Description: as for outcome 83
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
10^12 cells per liter
  Baseline, n=21 | 4.308 (0.3103)
  Day 21, n=17: number analyzed (Participants) | 17
  Day 21, n=17 | 4.356 (0.2518)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 4.383 (0.2998)

85. Secondary Outcome: Period 1: Absolute Values of Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter hematocrit. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Proportion of red blood cells in blood
  Baseline | 0.3783 (0.02759)
  Day 10 | 0.3769 (0.02467)

86. Secondary Outcome: Period 2: Absolute Values of Hematology Parameter: Hematocrit
Description: as for outcome 85
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Proportion of red blood cells in blood
  Baseline, n=21 | 0.3791 (0.02457)
  Day 21, n=17: number analyzed (Participants) | 17
  Day 21, n=17 | 0.3848 (0.02650)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 0.3895 (0.02969)

87. Secondary Outcome: Period 1: Absolute Values of Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time points for the analysis of hematology parameter hemoglobin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Grams per liter
  Baseline | 128.0 (10.06)
  Day 10 | 127.2 (9.29)

88. Secondary Outcome: Period 2: Absolute Values of Hematology Parameter: Hemoglobin
Description: as for outcome 87
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Grams per liter
  Baseline, n=21 | 128.5 (8.61)
  Day 21, n=17: number analyzed (Participants) | 17
  Day 21, n=17 | 129.5 (10.22)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 132.1 (11.23)

89. Secondary Outcome: Period 1: Absolute Values of Urine Concentration: Urine Specific Gravity
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Ratio
  Baseline | 1.0136 (0.00693)
  Day 10 | 1.0159 (0.00766)

90. Secondary Outcome: Period 2: Absolute Values of Urine Concentration: Urine Specific Gravity
Description: as for outcome 89
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Ratio
  Baseline, n=21 | 1.0162 (0.00792)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 1.0134 (0.00982)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 1.0139 (0.00807)

91. Secondary Outcome: Period 1: Absolute Values of Urine Concentration: Urine Urobilinogen
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Micromoles per liter
  Baseline | 3.3860 (0.00000)
  Day 10 | 5.1526 (4.66388)

92. Secondary Outcome: Period 2: Absolute Values of Urine Concentration: Urine Urobilinogen
Description: as for outcome 91
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Micromoles per liter
  Baseline, n=21 | 5.3209 (4.85645)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 7.9007 (6.56981)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 4.1827 (3.28490)

93. Secondary Outcome: Period 1: Absolute Values of Urine Concentration: Urine pH
Description: Urine samples were collected at indicated time points for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
pH
  Baseline | 6.09 (0.468)
  Day 10 | 5.87 (0.310)

94. Secondary Outcome: Period 2: Absolute Values of Urine Concentration: Urine pH
Description: as for outcome 93
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
pH
  Baseline, n=21 | 5.88 (0.312)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 6.28 (0.428)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 6.12 (0.219)

95. Secondary Outcome: Period 1: Number of Participants With Abnormal Urinalysis Parameters Using Dipstick Method.
Description: The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters (ketones, glucose, bilirubin, occult blood, nitrite and blood protein) can be read as positive, trace, 1+, 2+, 3+ and 4+ indicating proportional concentrations in the urine sample. Only participants with abnormal findings for urinalysis at any visit has been presented.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Participants
  Urine Ketone, Day 10, Trace | 1
  Urine Ketone, Day 10, 1+ | 1
  Urine leukocyte esterase, Day 10, 1+ | 2
  Urine Nitrite, Baseline, Positive | 1
  Urine occult blood, Baseline, 1+ | 1
  Urine occult blood, Baseline, 2+ | 2
  Urine occult blood, Baseline, 3+ | 2
  Urine occult blood, Day 10, Trace | 1
  Urine occult blood, Day 10, 1+ | 2
  Urine occult blood, Day 10, 3+ | 1
  Urine protein, Day 10, Trace | 1

96. Secondary Outcome: Period 2: Number of Participants With Abnormal Urinalysis Parameters Using Dipstick Method.
Description: as for outcome 95
Time Frame: Baseline (Day 10) and at Days 21 and 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Participants
  Urine Ketone, Baseline, Trace | 1
  Urine Ketone, Baseline, 1+: number analyzed (Participants) | 17
  Urine Ketone, Baseline, 1+ | 1
  Urine Ketone, Day 21, Trace: number analyzed (Participants) | 17
  Urine Ketone, Day 21, Trace | 1
  Urine Ketone, Day 24, 2+ | 1
  Urine leukocyte esterase, Baseline, 1+ | 2
  Urine leukocyte esterase, Day 21, 1+ | 1
  Urine Nitrite, Day 21, Positive | 1
  Urine Nitrite, Day 24, Positive | 1
  Urine occult blood, Baseline, Trace | 1
  Urine occult blood, Baseline, 1+ | 2
  Urine occult blood, Baseline, 3+ | 1
  Urine occult blood, Day 21, Trace | 3
  Urine occult blood, Day 21, 3+ | 1
  Urine occult blood, Day 24, Trace | 1
  Urine occult blood, Day 24, 1+ | 2
  Urine occult blood, Day 24, 2+ | 1
  Urine occult blood, Day 24, 3+ | 1
  Urine Protein, Baseline, Trace | 1

97. Secondary Outcome: Period 1: Absolute Values of ECG Mean Heart Rate
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure heart rate. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Beats per minute
  Baseline | 67.9 (10.09)
  Day 10 | 67.0 (7.07)

98. Secondary Outcome: Period 2: Absolute Values of ECG Mean Heart Rate
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure heart rate. Baseline is defined as the average of the triplicate predose assessments on Day 11.
Time Frame: Baseline (Day 11, Pre-dose) and at Day 11: 2, 4, 6 hours, Day 15: 2, 4, 6 hours, Day 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Beats per minute
  Baseline, n=21 | 64.6 (8.49)
  Day 11: 2 hours, n=21 | 67.4 (7.89)
  Day 11: 4 hours, n=21 | 64.0 (6.73)
  Day 11: 6 hours, n=21 | 71.3 (7.59)
  Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  Day 15: 2 hours, n=18 | 67.9 (9.42)
  Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  Day 15: 4 hours, n=18 | 65.8 (9.53)
  Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  Day 15: 6 hours, n=18 | 67.2 (8.80)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 67.8 (7.72)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 64.5 (7.41)

99. Secondary Outcome: Period 1: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF Interval, and QTcB Interval
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure PR interval, QRS duration, QT Interval, QTcF Interval and QTcB interval. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Milliseconds
  PR interval, Baseline | 156.1 (20.37)
  PR interval, Day 10 | 158.6 (19.93)
  QRS duration, Baseline | 85.7 (9.86)
  QRS duration, Day 10 | 85.9 (8.81)
  QT interval, Baseline | 389.8 (22.39)
  QT interval, Day 10 | 386.8 (19.95)
  QTcF interval, Baseline | 404.7 (13.56)
  QTcF interval, Day 10 | 400.6 (12.77)
  QTcB interval, Baseline | 412.0 (18.41)
  QTcB interval, Day 10 | 407.4 (14.28)

100. Secondary Outcome: Period 2: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF and QTcB Interval
Description: Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure PR Interval, QRS Duration, QT Interval, QTcF and QTcB Interval. Baseline is defined as the average of the triplicate predose assessments on Day 11.
Time Frame: Baseline (Day 11, Pre-dose) and at Day 11- 2, 4, 6 hours, Day 15- 2, 4, 6 hours, Day 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Milliseconds
  PR interval, Baseline, n=21 | 159.1 (18.22)
  PR interval, Day 11: 2 hours, n=21 | 159.4 (19.73)
  PR interval, Day 11: 4 hours, n=21 | 161.0 (18.73)
  PR interval, Day 11: 6 hours, n=21 | 157.2 (20.08)
  PR interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  PR interval, Day 15: 2 hours, n=18 | 158.7 (21.29)
  PR interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  PR interval, Day 15: 4 hours, n=18 | 159.8 (17.11)
  PR interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  PR interval, Day 15: 6 hours, n=18 | 158.1 (17.46)
  PR interval, Day 21, n=18: number analyzed (Participants) | 18
  PR interval, Day 21, n=18 | 162.1 (18.06)
  PR interval, Day 24, n=17: number analyzed (Participants) | 17
  PR interval, Day 24, n=17 | 162.8 (15.26)
  QRS duration, Baseline, n=21 | 85.5 (7.40)
  QRS duration, Day 11: 2 hours, n=21 | 83.3 (6.57)
  QRS duration, Day 11: 4 hours, n=21 | 84.9 (10.17)
  QRS duration, Day 11: 6 hours, n=21 | 85.2 (8.05)
  QRS duration, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QRS duration, Day 15: 2 hours, n=18 | 84.8 (6.68)
  QRS duration, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QRS duration, Day 15: 4 hours, n=18 | 84.6 (8.33)
  QRS duration, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QRS duration, Day 15: 6 hours, n=18 | 83.6 (8.44)
  QRS duration, Day 21, n=18: number analyzed (Participants) | 18
  QRS duration, Day 21, n=18 | 84.1 (9.46)
  QRS duration, Day 24, n=17: number analyzed (Participants) | 17
  QRS duration, Day 24, n=17 | 83.5 (8.60)
  QT interval, Baseline, n=21 | 394.2 (22.09)
  QT interval, Day 11: 2 hours, n=21 | 377.8 (20.18)
  QT interval, Day 11: 4 hours, n=21 | 396.5 (21.88)
  QT interval, Day 11: 6 hours, n=21 | 382.5 (22.01)
  QT interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QT interval, Day 15: 2 hours, n=18 | 382.9 (18.90)
  QT interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QT interval, Day 15: 4 hours, n=18 | 392.8 (24.36)
  QT interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QT interval, Day 15: 6 hours, n=18 | 395.3 (25.60)
  QT interval, Day 21, n=18: number analyzed (Participants) | 18
  QT interval, Day 21, n=18 | 385.7 (25.68)
  QT interval, Day 24, n=17: number analyzed (Participants) | 17
  QT interval, Day 24, n=17 | 394.2 (22.25)
  QTcF interval, Baseline, n=21 | 403.2 (12.93)
  QTcF interval, Day 11: 2 hours, n=21 | 391.8 (10.63)
  QTcF interval, Day 11: 4 hours, n=21 | 404.6 (12.78)
  QTcF interval, Day 11: 6 hours, n=21 | 404.5 (14.13)
  QTcF interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 15: 2 hours, n=18 | 398.2 (11.51)
  QTcF interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 15: 4 hours, n=18 | 403.6 (11.73)
  QTcF interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 15: 6 hours, n=18 | 409.3 (12.19)
  QTcF interval, Day 21, n=18: number analyzed (Participants) | 18
  QTcF interval, Day 21, n=18 | 400.8 (13.69)
  QTcF interval, Day 24, n=17: number analyzed (Participants) | 17
  QTcF interval, Day 24, n=17 | 403.0 (12.02)
  QTcB interval, Baseline, n=21 | 407.2 (16.45)
  QTcB interval, Day 11: 2 hours, n=21 | 398.7 (12.38)
  QTcB interval, Day 11: 4 hours, n=21 | 408.2 (12.46)
  QTcB interval, Day 11: 6 hours, n=21 | 415.4 (15.09)
  QTcB interval, Day 15: 2 hours, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 15: 2 hours, n=18 | 405.5 (16.82)
  QTcB interval, Day 15: 4 hours, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 15: 4 hours, n=18 | 408.8 (13.73)
  QTcB interval, Day 15: 6 hours, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 15: 6 hours, n=18 | 415.9 (11.36)
  QTcB interval, Day 21, n=18: number analyzed (Participants) | 18
  QTcB interval, Day 21, n=18 | 407.9 (11.29)
  QTcB interval, Day 24, n=17: number analyzed (Participants) | 17
  QTcB interval, Day 24, n=17 | 407.2 (12.99)

101. Secondary Outcome: Period 1: Absolute Values of Vital Signs: SBP and DBP
Description: SBP and DBP were assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline is defined as the average of the triplicate predose assessments on Day 11.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Millimeters of mercury
  SBP, Baseline | 115.7 (8.50)
  SBP, Day 10 | 111.4 (12.58)
  DBP, Baseline | 71.9 (8.87)
  DBP, Day 10 | 69.1 (8.71)

102. Secondary Outcome: Period 2: Absolute Values of Vital Signs: SBP and DBP
Description: SBP and DBP were assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Millimeters of mercury
  SBP, Baseline, n=21 | 110.0 (8.24)
  SBP, Day 15, n=19: number analyzed (Participants) | 19
  SBP, Day 15, n=19 | 113.3 (6.63)
  SBP, Day 21, n=18: number analyzed (Participants) | 18
  SBP, Day 21, n=18 | 110.1 (5.22)
  SBP, Day 24, n=17: number analyzed (Participants) | 17
  SBP, Day 24, n=17 | 114.5 (7.00)
  DBP, Baseline, n=21 | 64.6 (7.69)
  DBP, Day 15, n=19: number analyzed (Participants) | 19
  DBP, Day 15, n=19 | 66.7 (5.85)
  DBP, Day 21, n=18: number analyzed (Participants) | 18
  DBP, Day 21, n=18 | 67.4 (6.01)
  DBP, Day 24, n=17: number analyzed (Participants) | 17
  DBP, Day 24, n=17 | 69.7 (6.63)

103. Secondary Outcome: Period 1: Absolute Values of Pulse Rate
Description: Pulse rate was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Beats per minute
  Baseline | 70.1 (10.20)
  Day 10 | 70.0 (9.28)

104. Secondary Outcome: Period 2: Absolute Values of Pulse Rate
Description: as for outcome 103
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Beats per minute
  Baseline, n=21 | 69.2 (12.19)
  Day 15, n=19: number analyzed (Participants) | 19
  Day 15, n=19 | 73.5 (8.62)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 69.4 (7.11)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 68.4 (7.63)

105. Secondary Outcome: Period 1: Absolute Values of Respiratory Rate
Description: Respiratory rate was assessed indicated time-points. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Breaths per minute
  Baseline | 13.6 (2.56)
  Day 10 | 15.8 (2.33)

106. Secondary Outcome: Period 2: Absolute Values of Respiratory Rate
Description: as for outcome 105
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Breaths per minute
  Baseline, n=21 | 13.2 (2.41)
  Day 15, n=19: number analyzed (Participants) | 19
  Day 15, n=19 | 15.1 (2.93)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 14.1 (1.88)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 14.5 (2.60)

107. Secondary Outcome: Period 1: Absolute Values of Temperature
Description: Temperature was assessed at indicated time-points. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, within each treatment.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)
Number analyzed (Participants) | 23
Degree Celsius
  Baseline | 36.66 (0.487)
  Day 10 | 36.77 (0.335)

108. Secondary Outcome: Period 2: Absolute Values of Temperature
Description: as for outcome 107
Time Frame: Baseline (Day 11, Pre-dose) and at Days 15, 21 and 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
Number analyzed (Participants) | 21
Degree Celsius
  Baseline, n=21 | 36.60 (0.434)
  Day 15, n=19: number analyzed (Participants) | 19
  Day 15, n=19 | 36.75 (0.391)
  Day 21, n=18: number analyzed (Participants) | 18
  Day 21, n=18 | 36.59 (0.424)
  Day 24, n=17: number analyzed (Participants) | 17
  Day 24, n=17 | 36.82 (0.481)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from Day -3 to Day -1 in Run-in period and up to Day 25 in Treatment period.
Description: Non-serious AEs and SAEs were reported for the safety population which comprised of all participants who received at least one dose of study medication.
Arm/Group | Portia - Run-in Period (Day -3 to Day -1) | Portia (0.3 mg EE/ 0.15 mg LNG) | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 5/23 | 9/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Portia - Run-in Period (Day -3 to Day -1) (N=23) | Portia (0.3 mg EE/ 0.15 mg LNG) (N=23) | Portia (0.3 mg EE/ 0.15 mg LNG)+GSK3640254 (N=21)
Transaminases increased (Investigations) | 0 | 4 | 1
Headache (Nervous system disorders) | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03984825/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03984825/SAP_001.pdf